CLINICAL TRIAL: NCT03759002
Title: Association Between Mean Platelet Volume With Echocardiographic Indices and Carotid Intima Media Thickness in Children With End Stage Renal Disease.
Brief Title: Association of Mean Platelet Volume and Cardiovascular Disease in Children With End Stage Renal Disease.
Status: Completed | Type: Observational
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amin Abedini, Medical researcher, Isfahan University of Medical Sciences
Other Study IDs: 395723
Record Dates: First submitted 2018-11-22; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Cardiovascular Diseases; Carotid Intimal Media Thickness; Left Ventricular Hypertrophy; Mean Platelet Volume; End Stage Renal Disease; Hemodialysis Complication; Peritoneal Dialysis Complication; Children
MeSH Terms: conditions — Cardiovascular Diseases; Hypertrophy, Left Ventricular; Kidney Failure, Chronic | interventions — Diagnostic Imaging; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Children with end stage renal disease
  Interventions: Diagnostic Test: Imaging; Other: Blood sampling
- Controls: Healthy sex- and age adjusted children
  Interventions: Diagnostic Test: Imaging; Other: Blood sampling

INTERVENTIONS:
Diagnostic Test: Imaging — Imaging including Echocardiography for determining cardiac indices (ejection fraction, left ventricular mass index, strain rate, global longitudinal strain) and Doppler ultrasound for measuring carotid intima media thickness
Other: Blood sampling — Blood sampling will performed on all participants for measuring hematological parameters including MPV.

SUMMARY:
Cardiovascular disease (CVD) is the major risk factor for death in end stage renal diseases (ESRD). Approximately 80% of ESRD patients have some degrees of left ventricular abnormalities at initiation of dialysis. Carotid intima media thickness (CIMT) has been widely accepted as an useful marker to assess CVD in ESRD children. In addition, cardiac mechanics parameters are used to evaluate cardiac function more precisely. However, measuring CIMT and cardiac mechanics parameters are expensive and difficult to perform as a routine method. Mean platelet volume (MPV) is a hematological index which shows the size of platelets. Uremic state causes inflammatory condition that affects MPV. Previous studies on people with normal renal function have shown that this parameter can also have association with CVD. However the data in children with ESRD is scarce. The aim of this study is to find a simple hematologic marker to use regularly in ESRD children finding patients at risk of CVD. Therefore, we will investigate the relationship between mean platelet volume and CIMT and cardiac mechanic parameters in children with ESRD.

ELIGIBILITY:
Inclusion Criteria:

* Children under 18 years who have being dialyzed (hemodialysis or peritoneal dialysis) regularly more than 6 months, as case group.
* Age and gender matched healthy children who have been referred for routine medical examination.

Exclusion Criteria:

* Patients with uncontrolled hypertension (until being stabled)
* Patients on any kind of antithrombotic agents or NSAIDs
* Severe obesity
* Diabetes patients
* Patients with a past history of CVD or stroke in the last 6 months
* Passive smokers who contacted daily with high smokers in their houses
* Patients with known hematologic diseases or malignancies (such as Fanconi Anemia)
* Uncontrolled hypothyroid or hyperthyroid patients
* Patients with recent (in the last 4 weeks) catheter or exit -site infection.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients group will be selected from children who referred to a tertiary care center of pediatric nephrology diseases.
  Controls will be chosen from healthy volunteers who will be visited for medical routine examination in the hospital staff.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
MPV in patients and controls | 1 year after study beginning
  Comparing the mean of MPV in patients and controls.
Echocardiographic indices in patients and controls | 1.5 years after study beginning
  Comparing the means of echocardiographic indices in patients and controls
Carotid intima media thickness in patients and controls | 2 years after study beginning
  Comparing the mean of carotid intima media thickness in patients and controls
Correlation between MPV and ejection fraction | 1.5 years after study beginning
  Determining correlation between the value of MPV with ejection fraction in patients
Correlation between MPV and left ventricular mass index | 1.5 years after study beginning
  Determining correlation between the value of MPV with left ventricular mass index in patients
Correlation between MPV and strain rate | 1.5 years after study beginning
  Determining correlation between the value of MPV with strain rate in patients
Correlation between MPV and global longitudinal strain | 1.5 years after study beginning
  Determining correlation between the value of MPV with global longitudinal strain in patients
Correlation between MPV and carotid intima media thickness | 2 years after study beginning
  Determining correlation between the value of MPV with carotid intima media thickness in patients

SECONDARY OUTCOMES:
MPV and thrombotic events | 2 years after study beginning
  Comparing the values of MPV in patients with and without previous histories of thrombotic events including arteriovenous fistula thrombosis, cerebrovascular accident, deep venous thrombosis, and cerebrovascular accident

CONTACTS AND LOCATIONS:
Overall Officials: Alaleh Gheissari, M.D., Principal Investigator — Professor of pediatric nephrology